CLINICAL TRIAL: NCT06479083
Title: Interdisciplinary and Intersectoral Telemedicine Evaluation, Coordination and Treatment in the Rhine Main+ Parkinson's Network
Brief Title: Interdisciplinary + Intersectoral Telemedicine Evaluation, Coordination + Treatment in RhineMain+ Parkinson's Network
Acronym: INSPIRE-PNRM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Hochschule für Wirtschaft und Gesellschaft Ludwigshafen Institut für Management, Ökonomie und Versorgung im Gesundheitsbereich (Unknown); Katholische Hochschule Mainz Fachbereich Gesundheit und Pflege (Unknown); Universitätsklinikum Frankfurt Zentrum der Neurologie und Neurochirurgie (Unknown); Techniker Krankenkasse Landesvertretung Rheinland-Pfalz (Unknown); DAK-Gesundheit Landesvertretung Rheinland-Pfalz und Saarland (Unknown)
Responsible Party: Principal Investigator, Sergiu Groppa, Univ.-Prof. Dr. med. Dr. h.c. Sergiu Groppa, MBA, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 01NVF22107; 2024-17454 (Registry Identifier: Ethic commission RLP)
Record Dates: First submitted 2024-06-24; First posted 2024-06-27 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease, Advanced Practice Nurse, Telemedical, Interdisciplinary, cross-sector care networks and pathways.
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Study design: mixed-method approach; randomized study design. Planned intervention period: 12 months.
Who Masked: Participant, Care Provider
Masking Description: The participants are randomized into two groups: Interventional and control group. Neither APN nor the patients know in which group they belong until the first visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Other): New intervention form
  Interventions: Other: New Intervention form including
- control group. (Other): Standard treatment for Parkinson Disease
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: New Intervention form including — The central element of the new form of care is the implementation of a tele medical evaluation and coordination function, which controls individualized treatment processes within the network. The individualized evaluation and coordination of treatment paths is carried out within the already existing Parkinson's network RheinMain+ by a non-physician medical specialist (APN) specially trained for the indication Parkinson's disease.
  Arms: Interventional group
Other: Standard treatment — The standard treatment which all compulsory insured patients get.
  Arms: control group.

SUMMARY:
Project objective: To improve the health care of Parkinson's disease patients in the ParkinsonNetz RheinMain+.

Hypothesis: Through the interdisciplinary and cross- sectoral networking in a tele medical network and the coordinating function of an "advanced practice nurse" (APN) specially trained for Parkinson's disease, the process quality within the network is increased and the individual health status is positively influenced.

DETAILED DESCRIPTION:
To effectively influence the long-term course of Parkinson´s a synergistic application of an individualized therapy program, which is tailored specifically to the symptoms and disease stages, is needed. The central element of the new form of care is the implementation of a tele medical evaluation and coordination function, which controls individualized treatment processes within the network. The individualized evaluation and coordination of treatment paths is carried out within the already existing Parkinson's network RheinMain+ by a non-physician medical specialist (APN) specially trained for the indication Parkinson's disease. In-depth assessments of the individual disease situation of the patients will take place. Based on these assessments, an evidence-based and patient-centered treatment and care plan is developed. The treatment plans are monitored, controlled and evaluated by the APNs using audiovisual or tele medical communication. In addition, APNs are empowered to initiate treatment interventions necessary to implement clinical guidelines and standards, and to take charge of these interventions as part of delegation processes. The APNs ensure that patients are cared for in accordance with needs and guidelines in all areas of care. To this end, they offer, among other things, training in the handling of patients with Parkinson's disease for other professional groups involved in the treatment process and not only have the patients in mind, but also include relatives and the supporting team.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary Parkinson's syndrome (G20.-) or atypical Parkinson's syndrome (G23.-, according to the current diagnostic criteria of the Movement Disorder Society, including the criteria of at least bradykinesia and rigidity or resting tremor must be present)
* In the care regions of Hesse and Rhineland-Palatinate
* Ability to give consent present

Exclusion Criteria:

- Severe dementia

* Severe depression
* Psychoses or other psychiatric or medical comorbidities that could affect the smooth implementation of the study protocol (e.g.

tumor disease with limited life expectancy, need for dialysis, etc.)

* Drug or alcohol addiction
* Women who are pregnant or breastfeeding
* Simultaneous participation in another interventional treatment study
* Illiteracy or insufficient language skills

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1354 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Are there differences in the change in Parkinson's-specific quality of life after 12 months of observation between the intervention group and the controll group- operationalized by the PDQ-39 | duration of the intervention: 24 months
  Parkinson´s Disease Quetionnaire -39 - to measure the differences in the change in Parkinson's-specific quality of life after 12 months of observation between the intervention group and the control group

SECONDARY OUTCOMES:
Are there differences in the change in motor symptoms after 12 months of observation between the intervention group and the control group measured with the MDS-Unified Parkinson's Disease Rating Scale part III (MDS-UPDRS III) | duration of the intervention: 24 months
  MDS-UPDRS III- to measure the differences in the change in motor symptoms after 12 months of observation between the intervention group and the control group
Are there differences in the change in quality of life across diseases after 12 months of observation between the intervention and the control group measured with the European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-5L) | duration of the intervention: 24 months
  EQ-5D-5L- to measure the differences in the change in quality of life across diseases after 12 months of observation between the intervention group and the control group

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Universtity of Saarland, Campus Homburg, Dept. of Neurology, Homburg
  - INSPIRE-PNRM+ Neuroimaging Center (NIC) University Medical Center of the Johannes Gutenberg University Mainz, Mainz

IPD SHARING:
Plan to Share IPD: No